CLINICAL TRIAL: NCT03317509
Title: The Effect of High Frequency Repetitive Transcranial Magnetic Stimulation on Advancing Parkinson's Disease With Dysphagia
Brief Title: The Effect of High Frequency rTMS on Advancing Parkinson's Disease With Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMS on Parkinson dysphagia
Record Dates: First submitted 2017-10-07; First posted 2017-10-23 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Advanced Parkinson's With Dysphagia
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real rTMS (Active Comparator): Each patient received high frequency stimulation (25 HZ), with intensity of 80% of resting motor threshold detected from the hand motor area, with total 2000 pulses for each hemisphere for 10 consecutive sessions totally over period of 10 days
  Interventions: Procedure: repetitive transcranial magnetic (rTMS)
- Sham rTMS (Sham Comparator): Each patient received rTMS with the same pulse as the first group but with the coil placed perpendicular to the scalp.
  Interventions: Procedure: repetitive transcranial magnetic (rTMS)

INTERVENTIONS:
Procedure: repetitive transcranial magnetic (rTMS) — Real rTMS high frequency stimulation (25 HZ), with intensity of 80% of resting motor threshold detected from the hand motor area, with total 2000 pulses for each hemisphere for 10 consecutive sessions totally over period of 10 days. Sham rTMS is the same pulse as the first group but with the coil placed perpendicular to the scalp.

SUMMARY:
This study aims to assess the therapeutic role of rTMS on parkinson's patients with dysphagia. Thirty PD patients with dysphagia using UK bank criteria for PD will recruited from outpatient clinic in Assuit University. All patients were admitted at Neuropsychiatric Department, Assiut University Hospital/ Assiut, Egypt. Each patient fulfilled the inclusion criteria as spontaneous swallows should be identified clearly when patients cannot perform voluntary swallows using clinical examination test. The patients will be allocated randomly into two groups one of which will receive real sessions of high frequency rTMS (25 HZ), with intensity of 80% of resting motor threshold detected from the hand motor area, with total 2000 pulses for each hemisphere for 10 consecutive sessions totally over period of 10 days with repeated booster session every month during the period of follow up among three months. The other will receive sham sessions. All subjects will be followed up by selected clinical rating scales at different intervals pre session, post 10 sessions, and after one, two and three months.

DETAILED DESCRIPTION:
This study aims to assess the therapeutic role of repetitive transcranial magnetic (rTMS) on parkinson's patients with dysphagia. Thirty PD patients with dysphagia using UK bank criteria for PD will recruited from outpatient clinic in Assuit University. All patients were admitted at, Neuropsychiatric Department, Assiut University Hospital/ Assiut, Egypt. Each patient fulfilled the inclusion criteria as spontaneous swallows should be identified clearly when patients cannot perform voluntary swallows using clinical examination test. The patients will be allocated randomly into two groups using closed envelops one of which will receive real sessions of high frequency rTMS (25 HZ), with intensity of 80% of resting motor threshold detected from the hand motor area, with total 2000 pulses for each hemisphere for 10 consecutive sessions totally over period of 10 days with repeated booster session every month during the period of follow up among three months. the other will receive sham sessions. All subjects after receiving the rTMS will be followed up by selected clinical rating scales at different intervals Pre session, post 10 sessions, after one, two and three months.

ELIGIBILITY:
Inclusion Criteria:

* All parkinson's disease patients who were diagnosed according to UK bank criteria for PD, Aged 50-75 years, with dysphagia

Exclusion Criteria:

* History of repeated head injury
* History of repeated cerebrovascular strokes
* History of defined encephalitis
* Oculogyric crisis, supranuclear gaze palsy
* Family history of more than one relative
* History of drug intake as antipsychotics or MPTP exposure
* Severe dementia, (MMSE < 23), Severe depression (H- D) < severe dysautonomia
* Cerebellar signs
* Babiniski sign
* Strictly unilateral features after 3 years
* Hydrocephalus or intracranial lesion on neuroimaging
* We also excluded patients with intracranial metallic devices or with pacemakers or any other device.
* Patients who were unable to give informed Consent because of severe anesthesia or cognitive deficit were not included.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-16 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
changes in dysphagia severity measurement | Three months
  Dysphagia severity changes measured by Dysphagia Handicap Index (DHI)

SECONDARY OUTCOMES:
swallowing changes pre and post 10 sessions using | ten days
  Measurement of swallowing changes pre and post 10 sessions using video fluoroscopy (VFS).

CONTACTS AND LOCATIONS:
Overall Officials: Eman M Khedr, Principal Investigator — Professor of Neurology, Faculty of Medicine, Assiut University
Locations (1):
- Eman Khedr, Asyut, Assiut, Egypt, Egypt